CLINICAL TRIAL: NCT03062696
Title: A Pilot Study of Cognitive-Behavioral Therapy for Rumination Disorder (CBT-RD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Drexel University (Other)
Responsible Party: Principal Investigator, Jennifer Thomas, Co-Director, Eating Disorders Clinical and Research Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017P000283
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Rumination Disorder
MeSH Terms: conditions — Rumination Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (CBT-RD) (Experimental): There is only one arm in this study - all participants will be in the same arm, as all participants will receive CBT-RD. There is no control group.
  Interventions: Behavioral: CBT-RD

INTERVENTIONS:
Behavioral: CBT-RD — 5-8 sessions of cognitive behavioral therapy for rumination disorder (CBT-RD), held once per week in an outpatient setting.

SUMMARY:
The primary aim of this study is to pilot cognitive behavioral therapy (CBT-RD) for 10 individuals ages 10 and older who have rumination disorder

DETAILED DESCRIPTION:
Rumination disorder (RD; also known as "rumination syndrome") is characterized by the repeated regurgitation of food during or soon after eating, which typically occurs at least a few times per week, frequently daily, with subsequent re-chewing, re-swallowing, or spitting out of the regurgitated material. Diaphragmatic breathing is a widely used technique for rumination as a competing response to the abdominal wall contraction hypothesized to trigger regurgitation. However, the efficacy of diaphragmatic breathing remains unknown and has mainly been delivered simply through a one-session instruction with an occasional follow-up.

In the absence of evidence-based treatments for RD, Dr. Jennifer Thomas has contributed to the creation of a manualized treatment, Cognitive-Behavioral Therapy for Rumination Disorder (CBT-RD) informed by published case reports and currently in use at the Eating Disorders Clinical and Research Program (EDCRP) at Massachusetts General Hospital and the Psychological Services Center at Drexel University. CBT-RD targets the habitual contraction of the abdominal wall and preceding events through the use of habit reversal, using primarily diaphragmatic breathing as a competing response.

This study involves a phone screen to determine eligibility, followed by 5-8 sessions of CBT-RD (approximately 50 minutes each). A battery of questionnaires will be administered at pre-treatment, post-treatment, and 3-month follow-up intervals.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 or above
* Experience repeated regurgitation of food during or soon after eating, consistent with rumination disorder
* If applicable, have stable psychiatric medication for the past three months

Exclusion Criteria:

* Currently engage (in past three months) in any regular compensatory behaviors (e.g., self-induced vomiting, laxative/diuretic use)
* Current diagnosis of anorexia nervosa
* Acute suicide risk
* Are currently receiving psychological treatment for rumination disorder
* Co-morbid clinically significant psychological disorder that would require attention beyond the study treatment (e.g., psychotic disorder, substance dependence)
* Current pregnancy

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Pica, Avoidant/Restrictive Food Intake Disorder, Rumination Disorder Interview (PARDI) | Change from baseline to 3-month follow-up
  A semi-structured interview to assess pica, Avoidant/Restrictive Food Intake Disorder (ARFID), and/or rumination disorder diagnosis, severity, and symptoms. We will use the PARDI to assess frequency and severity of rumination behavior specifically.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Thomas, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Ani Keshishian, Boston, Massachusetts
  - Drexel University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No